CLINICAL TRIAL: NCT07139262
Title: Assessing the Impact of Climate-Resilient Disaster Preparedness Education on Nursing Students' Knowledge and Skills: A Quasi-Experimental Study at Jouf University, Saudi Arabia
Brief Title: Climate-Resilient Disaster Preparedness Education to Improve Knowledge and Skills in Nursing Students: A Quasi-Experimental Study
Acronym: CRDP-NurseEd
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mostafa Shaban, Lecturer, Jouf University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: KFSU-BC-A; KFU-IRB-2025-NUR-014 (Registry Identifier: Institutional Review Board (IRB) Number)
Record Dates: First submitted 2025-08-17; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Climate-Resilient Disaster Preparedness; Disaster Nursing Education; Emergency Preparedness in Nursing Students; Nursing Education - Climate Change and Disasters
Keywords: Nursing education; Disaster preparedness; Climate change; Emergency response training; Quasi-experimental study

STUDY DESIGN:
Intervention Model Description: A two-arm parallel quasi-experimental design was used. Participants were assigned to either the intervention group (climate-resilient disaster preparedness education) or the control group (usual curriculum).
Who Masked: Outcomes Assessor
Masking Description: Independent faculty assessors, who were not involved in delivering the intervention and unaware of group allocation, evaluated students' knowledge tests and OSCE checklists.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention - Climate-Resilient Disaster Preparedness Education (Experimental): Participants in this arm received a structured climate-resilient disaster preparedness education program developed for undergraduate nursing students. The program included four weekly sessions (2 hours each) delivered through lectures, interactive workshops, and simulation-based training. Content focused on disaster risk reduction, emergency response, climate-related hazards, triage, and resilience-building strategies. Educational materials were adapted to Saudi context and validated by experts.
  Interventions: Behavioral: Climate-Resilient Disaster Preparedness Education Program; Other: Standard Nursing Curriculum
- Control - Standard Nursing Curriculum (Active Comparator): Participants in this arm continued their regular nursing curriculum without additional training in disaster preparedness or climate resilience. They did not receive the specialized education sessions provided to the intervention group but were exposed to general nursing education as part of their academic program.
  Interventions: Behavioral: Climate-Resilient Disaster Preparedness Education Program; Other: Standard Nursing Curriculum

INTERVENTIONS:
Behavioral: Climate-Resilient Disaster Preparedness Education Program — A structured educational program designed to enhance nursing students' knowledge and skills in climate-resilient disaster preparedness. The program consisted of four weekly sessions (2 hours each) delivered through lectures, interactive group discussions, and simulation-based exercises. Core content included disaster risk reduction principles, emergency response protocols, climate-related hazard preparedness, psychological first aid, triage procedures, and resilience-building strategies. Training materials were validated by subject matter experts and culturally adapted for the Saudi nursing education context.
Other: Standard Nursing Curriculum — Participants continued their regular undergraduate nursing curriculum without additional specialized training in disaster preparedness or climate resilience. This curriculum provided foundational nursing education but did not include structured sessions on climate-related disaster management or resilience-building.

SUMMARY:
This study aims to evaluate the impact of a structured climate-resilient disaster preparedness education program on undergraduate nursing students' knowledge and practical skills. Climate change has intensified the frequency and severity of disasters, increasing the need for health professionals who are trained to respond effectively. Nursing students, as future frontline providers, must be equipped with both theoretical knowledge and hands-on competencies to manage disaster situations that are influenced by climate variability.

The study was conducted at Jouf University, Saudi Arabia, using a quasi-experimental design with intervention and control groups. A total of 160 undergraduate nursing students were recruited and randomly assigned at the class level (80 intervention, 80 control). The intervention group participated in a tailored disaster preparedness training program incorporating lectures, interactive workshops, and simulation-based exercises with a focus on climate-resilient responses. The control group continued with their standard nursing curriculum.

Outcomes were measured using validated instruments: a disaster preparedness knowledge questionnaire and an Objective Structured Clinical Examination (OSCE) for disaster management skills. Assessments were conducted at baseline, immediately post-intervention, and at a 4-week follow-up to evaluate retention.

The primary hypothesis is that students who receive the climate-resilient disaster preparedness education will demonstrate significantly greater improvement in knowledge and skills compared to those in the control group. Findings will provide evidence for integrating climate-resilient disaster preparedness into undergraduate nursing curricula to strengthen health workforce readiness for emerging global health challenges.

DETAILED DESCRIPTION:
Disasters linked to climate change pose a growing challenge to health systems worldwide, with increased frequency of extreme weather events, floods, heatwaves, and pandemics. Nurses are among the largest sector of the health workforce and play a pivotal role in disaster preparedness and response. However, traditional nursing curricula often lack structured training in climate-resilient disaster preparedness. Addressing this educational gap is critical for building a workforce capable of protecting public health in the face of climate variability.

This quasi-experimental study was conducted at Jouf University, Saudi Arabia, to assess the effect of climate-resilient disaster preparedness education on nursing students' knowledge and clinical skills. The study enrolled 160 undergraduate nursing students (80 assigned to the intervention arm, 80 to the control arm). After accounting for attrition, 78 students in the intervention group and 79 in the control group completed the study.

Intervention:

The intervention group received a structured disaster preparedness training program designed in alignment with World Health Organization (WHO) and International Council of Nurses (ICN) recommendations. The program consisted of:

Didactic sessions covering disaster types, climate-related risk factors, and preparedness principles.

Interactive workshops emphasizing risk assessment, triage, evacuation, and communication during disasters.

Simulation-based exercises using Objective Structured Clinical Examination (OSCE) stations to practice disaster response in scenarios such as floods, heat emergencies, and mass casualty incidents.

The program was delivered over a 4-week period, totaling 20 contact hours. Faculty members with expertise in disaster nursing and climate health facilitated the sessions.

Control Group:

The control group continued with the standard nursing curriculum without additional disaster-specific training during the study period.

Outcomes:

Primary Outcome: Change in disaster preparedness knowledge (measured by a validated questionnaire, developed by Alim et al., adapted and validated into Arabic).

Secondary Outcome: Change in disaster preparedness skills (measured through OSCE checklists developed by the WHO and validated for reliability in this context).

Additional Outcome: Retention of knowledge and skills at 4 weeks post-training.

Data Collection and Analysis:

Data were collected at three time points: baseline (pre-test), immediately after the intervention (post-test), and 4 weeks later (follow-up). Statistical analysis included paired t-tests to assess within-group changes, independent t-tests and ANCOVA for between-group differences, and calculation of effect sizes (Cohen's d).

Ethical Considerations:

The study was approved by the Jouf University Institutional Review Board (IRB No. KFU-IRB-2025-NUR-014). Written informed consent was obtained from all participants. Participation was voluntary, and confidentiality was maintained throughout.

Significance:

This study addresses a critical gap in nursing education by integrating climate-resilient disaster preparedness into the curriculum. The findings are expected to contribute evidence for policy-makers, educators, and accreditation bodies to strengthen disaster preparedness competencies in nursing programs, ultimately enhancing workforce readiness to respond to climate-related emergencies.

ELIGIBILITY:
Inclusion Criteria:

Undergraduate nursing students enrolled at Jouf University.

Aged between 18 and 30 years.

Registered in the second or third academic year at the time of study.

Willing to provide informed consent and participate voluntarily.

Able to attend all training sessions and complete pre-, post-, and follow-up assessments.

Exclusion Criteria:

Students who previously attended formal disaster preparedness or emergency management training outside the standard curriculum.

Students with physical or psychological conditions that may limit participation in simulation-based activities (e.g., mobility restrictions, severe anxiety disorders).

Final-year students due to scheduling conflicts with clinical placements.

Students who decline to provide written informed consent.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-08-20 (Estimated); Primary Completion 2025-09-18 (Estimated); Study Completion 2025-10-18 (Estimated)

PRIMARY OUTCOMES:
Change in Knowledge of Climate-Resilient Disaster Preparedness | Baseline (pre-test), immediately post-intervention, and 4-week follow-up
  Knowledge was measured using the Disaster Preparedness Knowledge

SECONDARY OUTCOMES:
Change in Disaster Preparedness Skills (OSCE Performance) | Baseline (pre-test), immediately post-intervention, and 4-week follow-up
  Practical disaster response skills were evaluated using a structured Objective

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the results reported in this study will be shared with other researchers upon reasonable request. Data will include demographic characteristics, pre- and post-test knowledge scores, skills (OSCE) scores, and follow-up outcomes.
Supporting Information: ICF

REFERENCES:
- [Background] Wade R. Climate Change and Healthcare: Creating a Sustainable and Climate-Resilient Health Delivery System. J Healthc Manag. 2023 Jul-Aug 01;68(4):227-238. doi: 10.1097/JHM-D-23-00096. PMID 37410987
- [Background] Rivero RM, Mittler R, Blumwald E, Zandalinas SI. Developing climate-resilient crops: improving plant tolerance to stress combination. Plant J. 2022 Jan;109(2):373-389. doi: 10.1111/tpj.15483. Epub 2021 Sep 22. PMID 34482588
- [Background] Chen X, Zhao C, Yun P, Yu M, Zhou M, Chen ZH, Shabala S. Climate-resilient crops: Lessons from xerophytes. Plant J. 2024 Mar;117(6):1815-1835. doi: 10.1111/tpj.16549. Epub 2023 Nov 15. PMID 37967090
- [Background] Romanello M, Napoli CD, Green C, Kennard H, Lampard P, Scamman D, Walawender M, Ali Z, Ameli N, Ayeb-Karlsson S, Beggs PJ, Belesova K, Berrang Ford L, Bowen K, Cai W, Callaghan M, Campbell-Lendrum D, Chambers J, Cross TJ, van Daalen KR, Dalin C, Dasandi N, Dasgupta S, Davies M, Dominguez-Salas P, Dubrow R, Ebi KL, Eckelman M, Ekins P, Freyberg C, Gasparyan O, Gordon-Strachan G, Graham H, Gunther SH, Hamilton I, Hang Y, Hanninen R, Hartinger S, He K, Heidecke J, Hess JJ, Hsu SC, Jamart L, Jankin S, Jay O, Kelman I, Kiesewetter G, Kinney P, Kniveton D, Kouznetsov R, Larosa F, Lee JKW, Lemke B, Liu Y, Liu Z, Lott M, Lotto Batista M, Lowe R, Odhiambo Sewe M, Martinez-Urtaza J, Maslin M, McAllister L, McMichael C, Mi Z, Milner J, Minor K, Minx JC, Mohajeri N, Momen NC, Moradi-Lakeh M, Morrissey K, Munzert S, Murray KA, Neville T, Nilsson M, Obradovich N, O'Hare MB, Oliveira C, Oreszczyn T, Otto M, Owfi F, Pearman O, Pega F, Pershing A, Rabbaniha M, Rickman J, Robinson EJZ, Rocklov J, Salas RN, Semenza JC, Sherman JD, Shumake-Guillemot J, Silbert G, Sofiev M, Springmann M, Stowell JD, Tabatabaei M, Taylor J, Thompson R, Tonne C, Treskova M, Trinanes JA, Wagner F, Warnecke L, Whitcombe H, Winning M, Wyns A, Yglesias-Gonzalez M, Zhang S, Zhang Y, Zhu Q, Gong P, Montgomery H, Costello A. The 2023 report of the Lancet Countdown on health and climate change: the imperative for a health-centred response in a world facing irreversible harms. Lancet. 2023 Dec 16;402(10419):2346-2394. doi: 10.1016/S0140-6736(23)01859-7. Epub 2023 Nov 14. PMID 37977174
- [Background] Ebi KL, Vanos J, Baldwin JW, Bell JE, Hondula DM, Errett NA, Hayes K, Reid CE, Saha S, Spector J, Berry P. Extreme Weather and Climate Change: Population Health and Health System Implications. Annu Rev Public Health. 2021 Apr 1;42:293-315. doi: 10.1146/annurev-publhealth-012420-105026. Epub 2021 Jan 6. PMID 33406378